CLINICAL TRIAL: NCT05895487
Title: Multicentered Observational Cohort Study on the Efficacy, Safety and Durability of the "UniLine" Epoxy-treated Prosthesis Made With Xenopericardium in the Treatment of Isolated Aortic and Mitral Valve Disease (UniLine RetroFit)
Brief Title: Study on Efficacy, Safety and Durability of the UniLine Prosthesis in the Treatment of Aortic and Mitral Valve Disease
Status: Recruiting | Type: Observational
Sponsor: Closed Joint-Stock Company NeoCor (Other)
Collaborators: CT Medical Limited Liability Company (Unknown); Research Institute for Complex Problems of Cardiovascular Diseases, Russia (Other)
Responsible Party: Sponsor
Other Study IDs: UL RF - 01
Record Dates: First submitted 2023-05-19; First posted 2023-06-08 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Diseases of Mitral and Aortic Valves; Rheumatic Disorders of Mitral and Aortic Valves; Other Congenital Malformations of Aortic and Mitral Valves; Valvular Heart Disease (Aortic and Mitral Valves); Mitral Valve Insufficiency and Aortic Valve Insufficiency
Keywords: acquired heart diseases; mitral valve; aortic valve; prosthetic heart valves; bioprosthetic valves "UniLine"; bioprosthetic valve dysfunction
MeSH Terms: conditions — Heart Valve Diseases; Mitral Valve Insufficiency; Aortic Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Acquired heart diseases continue to remain one of the most common causes of cardiac mortality and morbidity. In the Russian Federation, open surgery treatment of acquired valvular heart diseases (AVHD) is performed in more than 40 regions by specialists from 92 healthcare organizations.

Treating aortic or mitral valve disease using the "UniLine" biological prosthesis is expected to improve survival rates. Supposedly, in vivo the "UniLine" biological prosthesis will show optimal hemodynamic characteristics and high resistance to structural valve degeneration and infectious damage, thus lowering the risk of dysfunction. Moreover, the risk of repeated intervention due to dysfunction of the "UniLine" bioprosthesis should not exceed the risk of the primary implantation. Supposedly, in the case of dysfunction of "UniLine" bioprosthesis it would be possible to perform repeated replacement using valve-in-valve technique.

The aim of the study is to assess the effectiveness, safety, durability of the "UniLine" epoxy-treated prosthesis and the long-term outcome of the treatment of isolated mitral and aortic valve diseases using this prosthesis.

In accordance with the objectives and hypothesis, the following data will be analyzed: actuarial and linear survival rates (general and cardiac), non-lethal prosthesis-associated complications, prosthetic dysfunction and repeated interventions.

Moreover, in vivo hemodynamic parameters of the prosthesis will be assessed: the area of the effective opening surface, peak and mean gradient of pressure and blood flow velocity.

The study will be conducted at the Research Institute of Complex Issues of Cardiovascular Diseases. Study protocol received sponsorship approval and approval by Local Ethics Committee of the Research Institute and Research Coordinating Committee. The study will enroll patients who underwent isolated mitral or aortic valve replacement; transthoracic echocardiography will be conducted in all patients available for in-person visit.

DETAILED DESCRIPTION:
Acquired heart diseases continue to remain one of the most common causes of cardiac mortality and morbidity. In Russia, heart valve diseases account for 7 to 25% of all cardiovascular diseases, moreover, they rank third as the cause of heart failure. Prosthetic heart valves commonly used as an effective treatment of acquired valvular heart diseases (AVHD). In the Russian Federation, open surgery treatment of AVHD is performed in more than 40 regions by specialists from 92 healthcare organizations. Surgeries on heart valves, being high-tech care, most effectively prolong the life of patients. Timely treatment of the disease allows 75-95% of patients to return to an active lifestyle and work. The purpose of surgical interventions is to increase life expectancy and to improve the quality of life, which can be achieved via adequate changes in intracardiac hemodynamics and reverse remodeling in the postoperative period.

Bioprosthetic heart valves, unlike most mechanical valves, are characterized by high thromboresistance, optimal (similar to native) hemodynamics parameters and quietness; they improve the quality of life of patients and do not require anticoagulant therapy in the long-term postoperative period. Moreover, bioprosthetic valve dysfunction develops slowly (within a few months or years), meaning that there is time for further examination and preoperative preparation, and a patient's life can be saved.

The "UniLine" bioprosthesis is designed for mitral or aortic valve replacement. This medical device has been used in clinical practice since 2008. Manufacturing of the "UniLine" bioprosthesis involves novel and innovative technologies, including high-precision thickness measurement and laser cutting for the leaflets, which prevents the unfolding of collagen structure along the edge of the cut, and ensures maximum uniformity of the material used, preventing the development of fatigue-induced changes. Unique modeling of leaflets provides complete coaptation. Anticalcification treatment with aminophosphonates contributes to a significant decrease in calcium-binding capacity, which helps to reduce the risk of dysfunction. The absence of synthetic components in the bioprosthesis should reduce the likelihood of endocarditis. Xenopericardium is preserved by using the epoxide compound (diglycidyl ether of ethylene glycol) under low pressure. Each "UniLine" bioprosthesis is subject to mandatory preclinical hydrodynamic assessment in accordance with the National Standards of the Russian Federation (GOST 26997-2003 and GOST 52999-2008). The "UniLine" atrioventricular biological prosthesis is manufactured in standard sizes 26, 28, 30 and 32, the "UniLine" aortic biological prosthesis is manufactured in standard sizes 21, 23, 25.

Treating aortic or mitral valve disease using the "UniLine" biological prosthesis is expected to improve survival rates. Supposedly, in vivo the "UniLine" biological prosthesis will show optimal hemodynamic characteristics and high resistance to structural valve degeneration and infectious damage, thus lowering the risk of dysfunction. Moreover, the risk of repeated intervention due to dysfunction of the "UniLine" bioprosthesis should not exceed the risk of the primary implantation. Supposedly, in the case of dysfunction of "UniLine" bioprosthesis it would be possible to perform repeated replacement using valve-in-valve technique.

The aim of the study is to assess the effectiveness, safety, durability of the "UniLine" epoxy-treated prosthesis and the long-term outcome of the treatment of isolated mitral and aortic valve diseases using this prosthesis.

In accordance with the objectives and hypothesis, the following data will be analyzed: actuarial and linear survival rates (general and cardiac), non-lethal prosthesis-associated complications, prosthetic dysfunction and repeated interventions.

Moreover, in vivo hemodynamic parameters of the prosthesis will be assessed: the area of the effective opening surface, peak and mean gradient of pressure and blood flow velocity.

The study will be conducted at the Research Institute of Complex Issues of Cardiovascular Diseases. Study protocol received sponsorship approval and approval by Ethics Committee of the Research Institute and Research Coordinating Committee. The study will enroll 2000 patients who underwent isolated mitral or aortic valve replacement; transthoracic echocardiography will be conducted in all patients available for in-person visit.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes aged 18 years and older who underwent isolated mitral or aortic valve replacement using the "UniLine" bioprosthesis
* No prior heart valve replacement

Exclusion Criteria:

* The presence of a mechanical or biological prosthesis in another position
* Prior valve repair
* Aortic aneurysm repair (ascending aorta)
* Resection of a left ventricular aneurysm
* Patients with active cancer and patients with history of cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 years and older who underwent isolated mitral or aortic valve replacement.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Long-term safety and durability of the "UniLine" epoxy-treated prosthesis made with xenopericardium in the treatment of isolated mitral and aortic valve diseases | Up to 12 years from the moment of implantation
  Long-term safety of the "UniLine" epoxy-treated prosthesis made with xenopericardium in the treatment of isolated mitral and aortic valve diseases will be evaluated by the frequency of complications associated with the valve.
  Device safety is defined as the absence of severe adverse events associated with the device or procedure, assessed by the following clinical phenomena:
  1. Death
  2. Severe complications of the heart
  3. Life-threatening bleeding
  4. Any bioprosthesis-related dysfunction, migration, thrombosis or other complication requiring an open-heart surgery or repeated intervention.
  5. Myocardial infarction (or ACS) or progression of a chronic form of ischemia requiring percutaneous coronary intervention or coronary artery bypass grafting
  6. Access site complications
  7. Stroke
The long-term durability of the bioprosthesis will be evaluated by assessing the hemodynamic characteristics of the bioprosthetic valve (data obtained by echocardiography). | Up to 12 years from the moment of implantation
  1. Peak and mean gradient on the atrioventricular bioprosthesis (as provided by manufacturer manufacturer).
  2. The effective orifice area of the bioprosthesis (as provided by manufacturer manufacturer).

SECONDARY OUTCOMES:
Frequency of adverse events | Up to 12 years from the moment of implantation
  Frequency of adverse events
Frequency of severe adverse events | Up to 12 years from the moment of implantation
  Frequency of severe adverse events
Frequency of adverse events associated with the device | Up to 12 years from the moment of implantation
  Frequency of adverse events associated with the device
Frequency of adverse events associated with the procedure | Up to 12 years from the moment of implantation
  Frequency of adverse events associated with the procedure
The absence of all-cause mortality | Up to 12 years from the moment of implantation
  The absence of all-cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Bogachev-Prokofiev, MD, PhD, Principal Investigator — National Medical Research Center named after Academician E.N. Meshalkin; Alexey Evtushenko, MD, PhD, Principal Investigator — Research Institute for Complex Issues of Cardiovascular Diseases
Locations (1):
- Federal State Budgetary Scientific Institution "Research Institute for Complex Issues of Cardiovascilar Diseases", Kemerovo, Russia